CLINICAL TRIAL: NCT05876273
Title: Adaptive Motif-Based Control (AMBC): Pilot 1 - Neural Net Implementation of Automated Insulin Delivery
Brief Title: Neural-net Artificial Pancreas (NAP)
Acronym: NAP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Boris Kovatchev, PhD, Principal Investigator, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 230058; R01DK133148 (NIH)
Record Dates: First submitted 2023-03-24; First posted 2023-05-25 (Actual); Results first posted 2024-07-31 (Actual); Last update posted 2024-07-31 (Actual); Status verified 2024-07

CONDITIONS: Type1 Diabetes
Keywords: Artificial Pancreas (AP); Diabetes Mellitus, Type 1; Insulin Pump; Continuous Glucose Monitor (CGM); Model Predictive Control (MPC); Automated Insulin Delivery (AID); Adaptive Motif-based Control (AMBC)
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Intervention Model Description: Randomized crossover: Participants will be randomized to two groups differing by the order of controller use: Group A: NAP, followed by UMPC; Group B: UMPC, followed by NAP.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (2):
- NAP first, then UMPC (Experimental): Participants will use the Neural Net Artificial Pancreas (NAP) algorithm for 18 hours. Then switch to the University of Virginia Model-Predictive Control (UMPC) for 18 hours.
  Interventions: Device: Neural-net Artificial Pancreas; Device: University of Virginia Model Predictive Control
- UMPC first, then NAP (Experimental): Participants will use the UMPC for 18 hours, then switch to NAP for 18 hours.
  Interventions: Device: Neural-net Artificial Pancreas; Device: University of Virginia Model Predictive Control

INTERVENTIONS:
Device: Neural-net Artificial Pancreas — NAP is a neural-net implementation of the previously tested UMPC algorithm (below).
  Other Names: NAP
Device: University of Virginia Model Predictive Control — A previously tested artificial pancreas control algorithm, based on a differential-equation model of the human metabolic system in diabetes.
  Other Names: UMPC

SUMMARY:
This study is intended to assess a Neural-net Artificial Pancreas (NAP) implementation of an established AP controller - the University of Virginia Model Predictive Control Algorithm (UMPC). The health outcomes achieved on NAP will be compared to the health outcomes achieved on UMPC in a randomized crossover design. The investigators will consent up to 20 participants, ages ≥18.0, with a goal of completing 15 participants.

DETAILED DESCRIPTION:
The study will follow a randomized cross-over design assessing glycemic control on a Neural-net Artificial Pancreas (NAP), compared to the previously tested University of Virginia Model Predictive Control (UMPC) algorithm, in a supervised hotel setting:

The study will involve Tandem t:slim X2 Control-IQ (CIQ) users who will continue to use their CIQ systems, except during the hotel sessions, which will use the DiAs prototyping platform, connected to a Tandem t:AP research pump and a Dexcom G6 sensor, and implementing NAP or UMPC. The study sensor will be the same sensor used by CIQ - it will be disconnected from CIQ and connected to DiAs.

Following enrollment, one week of automated insulin delivery (AID) data will be downloaded from the participants' pumps or t:connect accounts and will be used to establish a baseline and initialize the control algorithms. Participants will be then studied at a local hotel for 20 hours, including an 18-hour experiment, randomly receiving either NAP or UMPC. Participants will then receive the opposite intervention either sequentially during the same hotel stay, or in a second hotel stay up to 28 days following the first hotel stay. During these 18-hour hotel sessions participants will be followed to compare blood glucose control on NAP vs. UMPC. The study meals and activities will be kept the same between study sessions.

The investigators will analyze non-inferiority of NAP compared to UMPC, but this pilot feasibility study is not powered to formally test noninferiority. The primary outcome is percent time in range (TIR) (70 to 180 mg/dL) on NAP vs UMPC. Secondary outcomes include frequency of hypoglycemia (time below range = TBR) and hyperglycemia (time above range = TAR), as well as other safety and control metrics.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥18.0 at time of consent.
2. Clinical diagnosis, based on investigator assessment, of type 1 diabetes for at least one year.
3. Currently using insulin for at least six months.
4. Currently using the Control-IQ automated insulin delivery system for at least one mont.
5. Hemoglobin A1c of ≤9%.
6. Using insulin parameters such as insulin to carb ratio and correction factor consistently in order to dose insulin for meals or corrections.
7. Access to internet and willingness to upload data during the study as needed.
8. If female of childbearing potential and sexually active, must agree to use a form of contraception to prevent pregnancy while a participant in the study. A negative serum or urine pregnancy test will be required for all females of childbearing potential within 24 hours prior to initiating the experimental algorithms. Participants who become pregnant will be discontinued from the study. Also, participants who during the study develop and express the intention to become pregnant within the timespan of the study will be discontinued.
9. Willingness to use the University of Virginia Diabetes Assistant system throughout study session.
10. Willingness to use personal Lispro (Humalog) or aspart (Novolog) during the study session.
11. Willingness not to start any new non-insulin glucose-lowering agent during the course of the trial (including Sodium-glucose cotransporter-2 inhibitors, metformin/biguanides, glucagon-like peptide-1 receptor agonists, Pramlintide, Dipeptidyl peptidase-4 inhibitors, Sulfonylureas and nutraceuticals).
12. Willingness to reschedule the hotel portion of the study if placed on systemic steroids (e.g. intravenous injection, intramuscular injection, intra-articular or oral routes).
13. An understanding and willingness to follow the protocol and signed informed consent.

Exclusion Criteria:

1. History of Diabetic Ketoacidosis (DKA) in the 12 months prior to enrollment.
2. Severe hypoglycemia resulting in seizure or loss of consciousness in the 12 months prior to enrollment.
3. Currently pregnant or intent to become pregnant during the trial.
4. Currently breastfeeding.
5. Currently being treated for a seizure disorder.
6. Treatment with Meglitinides/Sulfonylureas at the time of hotel study.
7. Use of metformin/biguanides, glucagon-like peptide-1 agonists, Pramlintide, Dipeptidyl peptidase-4 inhibitors, Sodium-glucose cotransporter-2 inhibitors, or nutraceuticals intended for glycemic control with a change in dose in the past month.
8. History of significant cardiac arrhythmia (except for benign premature atrial contractions and benign premature ventricular contractions which are permitted or previous ablation of arrhythmia without recurrence which may be permitted) or active cardiovascular disease.
9. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol such as the following examples:

   1. Inpatient psychiatric treatment in the past 6 months.
   2. Presence of a known adrenal disorder.
   3. Uncontrolled thyroid disease.
10. A known medical condition that in the judgment of the investigator might interfere with the completion of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2023-05-30 (Actual); Primary Completion 2023-09-08 (Actual); Study Completion 2023-09-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boris P Kovatchev, PhD, Study Director — University of Virginia Center for Diabetes Technology; Sue A Brown, MD, Principal Investigator — University of Virginia Center for Diabetes Technology
Locations (1):
- University of Virginia Center for Diabetes Technology, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
Will follow the NIH Data Sharing Policy and Implementation Guidance on sharing research resources for research purposes to qualified individuals in the scientific community.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Generally, data will be made available after the primary publications of each study.
Access Criteria: The Data Sharing Agreements will be formulated by the study team.

REFERENCES:
- [Result] Kovatchev B, Castillo A, Pryor E, Kollar LL, Barnett CL, DeBoer MD, Brown SA. Neural-Net Artificial Pancreas: A Randomized Crossover Trial of a First-in-Class Automated Insulin Delivery Algorithm. Diabetes Technol Ther. 2024 Jun;26(6):375-382. doi: 10.1089/dia.2023.0469. PMID 38277161
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/38277161/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study is intended to assess a Neural-net Artificial Pancreas (NAP) implementation of an established AP controller - the University of Virginia Model Predictive Control Algorithm (UMPC). The health outcomes achieved on NAP will be compared to the health outcomes achieved on UMPC in a randomized crossover design. The investigators will consent up to 20 participants, ages ≥18.0, with a goal of completing 15 participants.
Period: Overall Study
Arm/Group | NAP First, Then UMPC | UMPC First, Then NAP
Started | 8 | 7
Completed | 8 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Participants: Participants completed two consecutive 20-hour hotel sessions, receiving in random order either NAP or UMPC
Arm/Group | All Participants
Number analyzed (Participants) | 15
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 2
Age, Continuous [Mean (Full Range); unit: years] | 47.9 [27.6 to 67.9]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 5
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 15
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 13
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 15
Percent Time in Range (70-180 mg/dL) [Mean (Standard Deviation); unit: Percent of time between 70-180 mg/dl] | 69.3 (13.4)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Time-in-Range (TIR) on NAP Versus UMPC.
Description: The primary outcome is percent of time in 70 to 180 mg/dL range on NAP vs UMPC.
Time Frame: 36 hours (two 18-hour experiments)
Measure: Mean (Standard Deviation); unit: Percent of time between 70-180 mg/dl
Groups:
- Overall Study: All subjects randomized
Arm/Group | Overall Study
Number analyzed (Participants) | 15
Percent of time between 70-180 mg/dl
  Time in Range (NAP) | 86.08 (6.5)
  Time in Range (UMPC) | 87.25 (12.9)
Statistical Analysis 1: Comparison: Overall Study; Test type: Other — The statistical analysis included general linear models (GLM), with repeated measures (NAP vs UMPC) and a covariate the 1-hour average CGM level prior to initiating either controller. This covariate was used to compute the adjusted performance differences between NAP and UMPC. The data was analyzed using the GLM procedures of IBM SPSS 28.0; p = 0.2, GLM with Repeated Measures — 1-hour average CGM level prior to initiating either controller was included as a covariate in the analysis. This covariate was used to compute the adjusted performance differences between NAP and UMPC; General linear models (GLM), with repeated measures (NAP vs UMPC)

2. Secondary Outcome: Percent of Time in Hyperglycemia.
Description: Percent CGM readings above 180 mg/dL.
Time Frame: 36 hours (two 18-hour experiments)
Measure: Mean (Standard Deviation); unit: Percent of time above 180 mg/dl
Groups:
- Overall Study: All participants randomized
Arm/Group | Overall Study
Number analyzed (Participants) | 15
Percent of time above 180 mg/dl
  Percent CGM readings above 180 mg/dL (NAP) | 11.93 (6.4)
  Percent CGM readings above 180 mg/dL (UMPC) | 10.96 (13.1)

3. Secondary Outcome: Percent of Time in Hypoglycemia.
Description: Percent CGM readings below 70 mg/dL.
Time Frame: 36 hours (two 18-hour experiments)
Measure: Mean (Standard Deviation); unit: Percent of time below 70 mg/dl
Arm/Group | Overall Study
Number analyzed (Participants) | 15
Percent of time below 70 mg/dl
  Percent CGM readings below 70 mg/dL (NAP) | 1.88 (2.25)
  Percent CGM readings below 70 mg/dL (UMPC) | 1.79 (2.1)

4. Secondary Outcome: System Functionality
Description: The investigator will observe, record, and tabulate any system malfunctions requiring study team intervention.
Time Frame: 36 hours (two 18-hour experiments)
Measure: Number; unit: Number of reportable device malfunctions
Arm/Group | Overall Study
Number analyzed (Participants) | 15
Number of reportable device malfunctions | 0

5. Secondary Outcome: Participant Feedback
Description: The investigator will obtain qualitative feedback form the participants regarding system functionality.
Time Frame: 36 hours (two 18-hour experiments)
Population: Data were not collected
Arm/Group | Overall Study
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Adverse event data were collected while participants were enrolled in the study (approximately 2 months)
Arm/Group | NAP First, Then UMPC | UMPC First, Then NAP
All-Cause Mortality (participants affected / at risk) | 0/8 | 0/7
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/7
Other Adverse Events (participants affected / at risk) | 0/8 | 0/7

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT05876273/Prot_SAP_000.pdf
  • Informed Consent Form (2023-06-19): https://cdn.clinicaltrials.gov/large-docs/73/NCT05876273/ICF_002.pdf